CLINICAL TRIAL: NCT06015776
Title: PGC-1, Purines and the Postmenopausal Heart
Brief Title: Purinergic Signaling and the Postmenopausal Heart
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Robina Matyal, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000151/13
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diastolic Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Sex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Atrial tissue containing atrial myocytes is snap frozen in liquid nitrogen and stored.
  Serum samples are also collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men: Men who are undergoing cardiac surgery
  Interventions: Other: Gender
- Women: Women who are undergoing cardiac surgery
  Interventions: Other: Gender

INTERVENTIONS:
Other: Gender — Differences between men and women will be observed

SUMMARY:
There is an increased risk of diastolic heart failure in post menopausal women. Estrogen plays a positive role in regulating molecular pathways in heart remodeling. Such pathways may work through purinergic signaling and its downstream effects on the heart's mitochondrial metabolism and angiogenic response to stress. Loss of estrogen functionality in post menopausal women may account for the increased risk of diastolic heart failure. The investigators will explore said pathways using cardiac tissue obtained from patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death of women in the United States, accounting for around 1 of every 3 deaths. Estrogen deficiency, as seen in aging women or after oophorectomy, has been linked to loss of cardiovascular protection, typically seen during reproductive life. Up to half of women evaluated for myocardial ischemia have normal appearing coronary arteries. These women can develop heart failure with a preserved ejection fraction (termed HFpEF) for which the etiology is unclear. Hormonal replacement therapy (HRT) after menopause remains controversial but current evidence cannot support this for either primary or secondary prevention of CVD. There are clearly modulatory influences on estrogenic signaling, that could well influence cardiovascular health in later life. Previous studies have demonstrated that estrogen improves energy production within the heart by increasing 5' adenosine monophosphate-activated protein (AMPK) and mitochondrial biogenesis via upregulation of peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α); a master switch of mitochondrial function, linked to vascular integrity and angiogenesis. Estrogen has been also found to modulate purinergic signaling by boosting expression of adenosine receptors and of CD39, the dominant endothelial ecto-ADPase that generates adenosine. There are also close relationships between purinergic signaling and dipeptidyl peptidase-4 (DPP-4; otherwise known as adenosine deaminase complexing protein 2 or CD26), possibly mediated by adenosine deaminase bioactivity. Decreased PGC-1α and aberrant purinergic signaling in metabolic syndrome may lead to impaired mitochondrial function, provoking diastolic dysfunction, and also result in impaired angiogenesis. The investigators hypothesize there are central roles of PGC-1α, purines and DPP-4 linked neuropeptide pathways in the control of angiogenesis and mitochondrial activity. These become increasingly disordered in setting of estrogen loss provoking development of metabolic syndrome, thereby exacerbating HFpEF and microvascular disease. Specific Aim 1: To determine how ischemia and cardiometabolic dysfunction in women's heart disease are exacerbated by the loss of puringeric pathways from estrogen deficiency. The investigators expect to determine that diastolic dysfunction is a functional consequence of this microvascular loss and cardiometabolic dessynchrony. Specific Aim 2: To evaluate the role of adenosingergic receptor activation and DPPIV inhibition on angiogenesis in a ovariectomized swine model of chronic myocardial ischemia and metabolic syndrome. Here, the investigators will explore relationships between the regulated and linkages in the exocytosis of nucleotides and neuropeptides, formation of nucleosides (adenosine) and alterations in angiogenic activity secondary to these. Summary: The investigators will study fundamental mechanisms in heart disease underpinning biological differences in women. The investigators will also offer new therapeutic strategies that target cardiac metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery under cardiopulmonary bypass.

Exclusion Criteria:

* Refusal to participate
* Emergency surgery
* Pre-existing heart block
* Preexisting atrial fibrillation
* Redo surgery
* Estrogen or hormone replacement therapy
* History of chronic heart failure
* History of major kidney disease

Ages: 30 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for elective cardiac surgery. Patients will be enrolled and consented during hospital admission for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparative quantification of expression of CD39 and adenosinergic receptors | 6 months
  Expression of CD39, ADORA2A and ADORA2B in cardiac tissue measured using Western blotting
Comparative quantification of expression of PGC-1 alpha, mitochondrial markers | 6 months
  Expression of PGC-1 alpha, AMPK and mitochondrial markers using Western blot
Comparative quantification of expression of angiogenic markers | 6 months
  Expression of angiogenic markers (PDGF, VEGF, Angiostatin)

CONTACTS AND LOCATIONS:
Overall Officials: Robina Matyal, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Professor of Anesthesia; Simon Robson, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center,Vice Chair Research
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No